CLINICAL TRIAL: NCT04457258
Title: PET Biodistribution Study of 68Ga-FAPI-46 in Patients With Sarcoma: An Exploratory Biodistribution Study With Histopathology Validation
Brief Title: 68Ga-FAPi-46 PET/CT Scan in Imaging Patients With Sarcoma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-000623; NCI-2020-03767 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-000623 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Sarcoma; Recurrent Sarcoma; Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — FAPI-46; Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (68Ga-FAPI-46 PET/CT) (Experimental): Patients receive 68Ga-FAPi-46 intravenously (IV), and then undergo PET/computed tomography (CT) over 20-90 minutes. On another day, patients receive 18F-FDG and then undergo PET/computed tomography (CT) according to standard of care procedures (if applicable).
  Interventions: Procedure: Computed Tomography; Drug: Gallium Ga 68 FAPi-46; Procedure: Positron Emission Tomography; Radiation: 18F-FDG

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Gallium Ga 68 FAPi-46 — Given IV
  Other Names: 68Ga-FAPi-46; Gallium-68-FAPi-46
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Radiation: 18F-FDG — Given IV
  Other Names: 18F-fluorodeoxyglucose

SUMMARY:
This early phase I trial studies an imaging technique called 68Ga-FAPi-46 PET/CT to determine where and to which degree the FAPI tracer (68Ga-FAPi-46) accumulates in normal and cancer tissues in patients with sarcoma. PET is an established imaging technique that utilizes small amounts of radioactivity attached to very minimal amounts of tracer, in the case of this research, 68Ga-FAPi. Because some cancers take up 68Ga-FAPi it can be seen with PET. CT utilizes x-rays that traverse body from the outside. CT images provide an exact outline of organs and potential inflammatory tissue where it occurs in patient's body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To define the biodistribution of gallium Ga 68 fibroblast activation protein inhibitor (FAPi)-46 (68Ga-FAPi-46) in normal and cancer tissues of patients with sarcoma with histopathology validation.

SECONDARY OBJECTIVES:

I. To evaluate whether 68Ga-FAPi-46 accumulation observed by positron emission tomography (PET) reflects geography, extent and degree of FAP expression determined by immuno-histochemistry (IHC).

II. To assess the 68Ga-FAPI-46 biodistribution correlation with fludeoxyglucose F-18 (18F-FDG) biodistribution and to define the frequency of the following phenotypes (FAP positive [+]/ FDG+, FAP negative [-]/ FDG+, FAP+/ FDG-, FAP-/ FDG-).

III. 3. To determine FAP expression profile and identify activating and loss of function mutations and gene rearrangement in available tumor tissue samples from patients with localized or metastatic sarcoma using RNA sequencing

OUTLINE:

Patients receive 68Ga-FAPi-46 intravenously (IV), and then undergo PET/computed tomography (CT) over 20-90 minutes. On another day, patients receive 18F-FDG and then undergo PET/computed tomography (CT) according to standard of care procedures (if applicable).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo surgical excision or biopsy of a suspected sarcoma primary, or a suspected recurrent or metastatic lesion.
* Patients who are ≥ 18 years old at the time of the radiotracer administration.
* Patients who can provide written informed consent.
* Patients who are able to remain still for duration of imaging procedures (up to one hour for each).

Exclusion Criteria:

* Patient is pregnant or nursing.
* Patients with any new cancer therapy between the baseline 18F-FDG PET/CT and the investigational FAPI PET/CT
* Patient has underlying disease which, based on the judgment of the investigator, might interfere with the collection of high quality data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-21 (Estimated)

PRIMARY OUTCOMES:
Biodistribution of gallium Ga 68 fibroblast activation protein inhibitor (FAPi)-46 (68Ga-FAPi-46) in normal and cancer tissues | At 20-90 minutes after injection
  Will be quantified by mean and maximum standardized uptake values (SUVmean and SUVmax).

SECONDARY OUTCOMES:
68Ga-FAPi-46 accumulation observed by positron emission tomography (PET)/computed tomography (CT) | Up to year 2
  Will be correlated with and validated by FAP expression in surgically removed or biopsy derived tumor tissue.
Frequency of the following phenotypes (FAP positive [+]/ fludeoxyglucose [FDG]+, FAP negative [-]/ FDG+, FAP+/ FDG-, FAP-/ FDG-) | Up to year 2
  To assess the 68Ga-FAPI-46 biodistribution correlation with 18F-FDG biodistribution and to define the frequency of the following phenotypes (FAP+/ FDG+, FAP-/ FDG+, FAP+/ FDG-, FAP-/ FDG-)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Calais, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States